CLINICAL TRIAL: NCT03801824
Title: Investigating the Effectiveness of a Low Glycemic Index on Glycemic Control and Pregnancy Outcomes in Women With Gestational Diabetes Mellitus: A Randomised Controlled Trial
Brief Title: Effect of Low Glycemic Index on Gestational Diabetes Mellitus
Acronym: MyLGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Barakatun Nisak Bt Mohd Yusof, Associate Professor, Universiti Putra Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 5450647
Record Dates: First submitted 2018-11-04; First posted 2019-01-14 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational Diabetes Mellitus; Glycemic index; Metabolic Response; Pregnancy Outcomes; Glycemic control
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Nutrition Therapy (Active Comparator): Subjects in this group receive a standard nutrition therapy based on local guidelines that is usually high in fibre with moderate to high glycemic index food
  Interventions: Other: Standard Nutrition Therapy
- Low Glycemic Index (Experimental): Subjects in this group receive intervention on low glycemic index foods
  Interventions: Other: Low Glycemic Index

INTERVENTIONS:
Other: Standard Nutrition Therapy — Subjects will be advised on standard diet appropriate for the management of Gestational Diabetes Mellitus (GDM) designed to be high in fiber and have moderate to high dietary glycemic index
  Arms: Standard Nutrition Therapy
Other: Low Glycemic Index — Subjects will be advised to eat low glycemic index foods
  Arms: Low Glycemic Index

SUMMARY:
The purpose of this study is to determine whether glycemic index is effective in the treatment of maternal glycemia and pregnancy outcomes in women with Gestational Diabetes Mellitus.

DETAILED DESCRIPTION:
1. This research is divided into 2, that are study I and study II

1. Study I, is to determine the long-term effects of intervention (low GI and SNT) on maternal glycemia, pregnancy outcomes and postprandial metabolic markers in women with GDM

   * A total of 110 women with confirmed diagnosis of GDM will be recruited
   * They will be randomized either to receive low GI (n=55) or Standard Nutrition Therapy (SNT; n=55)
   * The intervention will be started as soon as the women being diagnosed with GDM and they will be followed-up every month until delivery and up to the 3-month postpartum.
   * The primary outcome measures include glycemic control parameters as assessed by fasting and postprandial glycemia, fructosamine, HbA1c, insulin level and requirement for insulin treatment.
   * Secondary outcomes include lipid profile, weight gain, measures of postprandial metabolic response (free fatty acid and triglyceride), pregnancy outcomes, and overall improvement in postpartum metabolic parameters.
2. Study II, a sub-Mixed-meal Tolerant Test (MTT) study will be conducted to determine postprandial glycemic and metabolic responses before and after 4-weeks of intensive intervention

   * During the 4-weeks of intensive intervention, the subjects will receive individualise counseling and daily food supply regarding the allocated study group.
   * A minimum of 19 subjects from a pool of 110 subjects who is participated in the intervention study will be recruited.
   * The MTT procedure is similar to the oral glucose tolerant test (OGTT) but the subject will be asked to consume the real mixed meals representing low and high GI foods rather than oral glucose solution.
   * Subject will be asked to consume the test meal (either low or high GI foods) and the blood will be sampled before and after consuming the test meal in two different occasions with 1-week wash-out period.
   * After one month of intensive intervention, 19 subjects from each arm will undergo the final HGI meal tolerant test (MTT3) and the same procedure of MTT 1 and 2
   * Approximately 32μl of capillary blood by finger-prick will be obtained 7 times per MTT session, which is every 30 minutes thereafter to complete 3-h postprandial meal for each set of meal tests.

ELIGIBILITY:
Study I

Inclusion Criteria:

* Pregnant women, aged 18-45 years
* Women diagnosed with Gestational Diabetes Mellitus (GDM) as early as 13 up to 28 weeks of gestation
* Pre-pregnancy BMI >23kg/m2 (using BMI cut-off point) for underweight and overweight of Asian as defined by World Health Organization (WHO, 2000)
* Treated with diet controlled or on insulin therapy
* Willing and able to comply with the study protocol

Exclusion Criteria:

* Any gastrointestinal disease that interferes with bowel function and nutritional intake (i.e., diabetes-related constipation or diarrhea secondary to neuropathy, diarrhea due to chronic inflammatory bowel disease, gastroparesis, gastrectomy, galactosemia, hyperemesis
* Any medical problem that requires steroid (i.e., arthritis, asthma, autoimmune diseases and skin conditions such as eczema
* Incapability to comply with study protocol or investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements

Study II

Inclusion Criteria:

* Pregnant women, aged 18-45 years
* Only women diagnosed with Gestational Diabetes Mellitus (GDM) between 16 and 28 weeks of gestation
* Pre-pregnancy BMI >23kg/m2 (using BMI cut-off point) for underweight and overweight of Asian as defined by WHO (2000)
* Treated with diet-controlled alone
* Hemoglobin ≥10mmol/l (WHO, 2011)
* Willing and able to comply with the protocol

Exclusion Criteria:

* Any gastrointestinal disease that interferes with bowel function and nutritional intake (i.e., diabetes-related constipation or diarrhea secondary to neuropathy, diarrhea due to chronic inflammatory bowel disease, gastroparesis, gastrectomy, galactosemia, hyperemesis)
* Currently on insulin therapy
* With known food allergy/ on a particular dietary requirement
* Incapability to comply with study protocol or investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Post meal blood glucose level | 12 weeks
  Average blood glucose profiles after breakfast, lunch and dinner measured using capillary blood glucose at home

SECONDARY OUTCOMES:
Level of Triglycerides | 12 weeks
  Changes in Fasting Triglycerides
Level of glycemic control | 4 weeks
  Changes in Fructosamine
Maternal weight gain | 12 weeks
  Changes in total weight gain based on Institute of Medicine (IOM) recommendations

OTHER OUTCOMES:
Level of post-meal blood glucose | 3 hour post-prandial
  Changes in post-meal blood glucose level

CONTACTS AND LOCATIONS:
Overall Officials: Barakatun-Nisak Mohd Yusof, PhD, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Cheras, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Louie JC, Markovic TP, Ross GP, Foote D, Brand-Miller JC. Timing of peak blood glucose after breakfast meals of different glycemic index in women with gestational diabetes. Nutrients. 2012 Dec 21;5(1):1-9. doi: 10.3390/nu5010001. PMID 23344248
- [Background] Moses RG, Barker M, Winter M, Petocz P, Brand-Miller JC. Can a low-glycemic index diet reduce the need for insulin in gestational diabetes mellitus? A randomized trial. Diabetes Care. 2009 Jun;32(6):996-1000. doi: 10.2337/dc09-0007. Epub 2009 Mar 11. PMID 19279301
- [Background] Grant SM, Wolever TM, O'Connor DL, Nisenbaum R, Josse RG. Effect of a low glycaemic index diet on blood glucose in women with gestational hyperglycaemia. Diabetes Res Clin Pract. 2011 Jan;91(1):15-22. doi: 10.1016/j.diabres.2010.09.002. Epub 2010 Nov 20. PMID 21094553
- [Background] Moses RG, Luebcke M, Davis WS, Coleman KJ, Tapsell LC, Petocz P, Brand-Miller JC. Effect of a low-glycemic-index diet during pregnancy on obstetric outcomes. Am J Clin Nutr. 2006 Oct;84(4):807-12. doi: 10.1093/ajcn/84.4.807. PMID 17023707
- [Background] Perichart-Perera O, Balas-Nakash M, Rodriguez-Cano A, Legorreta-Legorreta J, Parra-Covarrubias A, Vadillo-Ortega F. Low Glycemic Index Carbohydrates versus All Types of Carbohydrates for Treating Diabetes in Pregnancy: A Randomized Clinical Trial to Evaluate the Effect of Glycemic Control. Int J Endocrinol. 2012;2012:296017. doi: 10.1155/2012/296017. Epub 2012 Nov 29. PMID 23251152